CLINICAL TRIAL: NCT02774798
Title: Correlation of Anal Acoustic Reflectometry Parameters With Degree of Rectal Intussusception and Prolapse
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016GA004
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Pelvic Floor Disorders
Keywords: Rectal Prolapse; Rectal Intussuception
MeSH Terms: conditions — Pelvic Floor Disorders; Rectal Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rectal Intussusception and Prolapse: AAR measurements will be taken from patients with suspected intra-rectal intussusception or rectal prolapse. Subgroup analysis will be performed after grading of rectal prolapse according to the Oxford Grading system. The subgroups will be:
  1. Oxford Grades 1 & 2 - intra-rectal intussusception
  2. Oxford Grades 3 & 4 - intra-anal intussusception
  3. Oxford grade 5 - Overt Rectal Prolapse

SUMMARY:
Anal Acoustic Reflectometry (AAR) is a reliable and reproducible technique that has been studied in our department over the last 6 years. Sound waves pass into a balloon placed in the anal canal and are used to measure the cross-sectional area. By gradually increasing and decreasing the pressure in the balloon the investigators can measure the pressure at which the cross-sectional area starts to increase and decrease, and the anal canal starts to open and close. This assessment mimics the natural opening and closing of the anal canal and the effect of squeezing the muscles.

Rectal intussusception occurs when the rectal wall telescopes into itself distally and is termed prolapse when it protrudes through the anal canal. Not all patients will require surgery and, for some, it can lead to debilitating symptoms of constipation, pain and faecal incontinence. Currently, the Oxford grading system through radiological testing is used for classifying severity of rectal intussusception and prolapse; however this does not give us sufficient information about the anal sphincter muscles.

The gold standard investigation of the anal sphincter muscles has been manometry which measures anal canal pressure at rest and during squeeze. However, it has limitations. In previous studies AAR has shown promise in the assessment of faecal incontinence and, that unlike manometry, it has been able to distinguish between different types of incontinence. Thus far, it has not been studied in patients with rectal intussusception and it is hoped that AAR parameters may provide an indication of when rectal intussusception becomes overt rectal prolapse. This can inform the clinician to guide further management of a group of patients with a condition that can have significant impact on quality of life.

DETAILED DESCRIPTION:
This an observational study based on not intervention. Patients are grouped depending on grade of prolapse, and all undergo the routine AAR investigation. Patients are grouped solely on differences in pathology already present and not on any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* Have capacity to consent to the study
* Patients with pelvic floor dysfunction and symptoms of rectal intussusception and rectal prolapse

Exclusion Criteria:

* Minors under the age of 18 years old
* Patients who lack capacity to consent
* Patients without pelvic floor dysfunction or symptoms of rectal intussusception or rectal prolapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the pelvic floor clinic and neurogastroenterology with symptoms of rectal prolapse
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Telford, Study Chair — University Hospital of South Manchester
Locations (1):
- University Hospital of South Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared. The correlations will be made with grade of oxford prolapse and then be grouped

REFERENCES:
- [Background] Klarskov N, Saaby ML, Lose G. A faster urethral pressure reflectometry technique for evaluating the squeezing function. Scand J Urol. 2013 Dec;47(6):529-33. doi: 10.3109/21681805.2013.776629. Epub 2013 Mar 19. PMID 23506115
- [Background] Hornung BR, Mitchell PJ, Carlson GL, Klarskov N, Lose G, Kiff ES. Comparative study of anal acoustic reflectometry and anal manometry in the assessment of faecal incontinence. Br J Surg. 2012 Dec;99(12):1718-24. doi: 10.1002/bjs.8943. PMID 23132420
- [Background] Mitchell PJ, Klarskov N, Telford KJ, Hosker GL, Lose G, Kiff ES. Viscoelastic assessment of anal canal function using acoustic reflectometry: a clinically useful technique. Dis Colon Rectum. 2012 Feb;55(2):211-7. doi: 10.1097/DCR.0b013e31823b2499. PMID 22228166
- [Background] Mitchell PJ, Klarskov N, Telford KJ, Hosker GL, Lose G, Kiff ES. Anal acoustic reflectometry: a new reproducible technique providing physiological assessment of anal sphincter function. Dis Colon Rectum. 2011 Sep;54(9):1122-8. doi: 10.1097/DCR.0b013e318223fbcb. PMID 21825892
- [Background] Collinson R, Cunningham C, D'Costa H, Lindsey I. Rectal intussusception and unexplained faecal incontinence: findings of a proctographic study. Colorectal Dis. 2009 Jan;11(1):77-83. doi: 10.1111/j.1463-1318.2008.01539.x. Epub 2008 Apr 28. PMID 18462221

RESULTS

PARTICIPANT FLOW:
Groups:
- Intra-rectal Intussusception (Oxford Groups 1 &2); Intra-anal Intussusception (Oxford Grades 3 & 4); Overt Rectal Prolapse (Oxford Grade 5): Patients grade of rectal prolapse depending on Oxford grading criteria
Period: Overall Study
Arm/Group | Intra-rectal Intussusception (Oxford Groups 1 &2) | Intra-anal Intussusception (Oxford Grades 3 & 4) | Overt Rectal Prolapse (Oxford Grade 5)
Started | 7 | 17 | 7
Completed | 7 | 17 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overt Rectal Prolapse (Oxford Garde 5): Patients grade of rectal prolapse depending on Oxford grading criteriaProlapse
- Total: Total of all reporting groups
Arm/Group | Intra-rectal Intussusception (Oxford Groups 1 &2) | Intra-anal Intussusception (Oxford Grades 3 & 4) | Overt Rectal Prolapse (Oxford Garde 5) | Total
Number analyzed (Participants) | 7 | 17 | 7 | 31
Age, Continuous [Median (Full Range); unit: years] | 53 [35 to 95] | 64 [35 to 70] | 68 [41 to 95] | 61 [35 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 6 | 26
  Male | 0 | 4 | 1 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 17 | 7 | 31

OUTCOME MEASURES:

1. Primary Outcome: Opening Pressure
Description: The pressure (in cmH20) at which the anal canl just begins to open
Time Frame: at specific time point of measurement up to 1 hour
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Intra-rectal Intussusception (Oxford Groups 1 &2) | Intra-anal Intussusception (Oxford Grades 3 & 4) | Overt Rectal Prolapse (Oxford Grade 5)
Number analyzed (Participants) | 7 | 17 | 7
cmH20 | 56.35 (16.64) | 39.01 (18.02) | 23.42 (14.52)

2. Secondary Outcome: Opening Elastance
Description: in cmH20/mm2 - the resistance of the anal canal to stretch
Time Frame: at specific time point of measurement up to 1 hour
Measure: Mean (Standard Deviation); unit: cmH20/mm2
Arm/Group | Intra-rectal Intussusception (Oxford Groups 1 &2) | Intra-anal Intussusception (Oxford Grades 3 & 4) | Overt Rectal Prolapse (Oxford Grade 5)
Number analyzed (Participants) | 7 | 17 | 7
cmH20/mm2 | 1.72 (7.82) | 1.19 (0.40) | 0.93 (0.34)

3. Secondary Outcome: Closing Pressure
Description: The pressure (cmH20) at whihc the anal canal just closes
Time Frame: at specific time point of measurement up to 1 hour
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Intra-rectal Intussusception (Oxford Groups 1 &2) | Intra-anal Intussusception (Oxford Grades 3 & 4) | Overt Rectal Prolapse (Oxford Grade 5)
Number analyzed (Participants) | 7 | 17 | 7
cmH20 | 33.31 (10.84) | 22.78 (12.53) | 13.58 (9.80)

4. Secondary Outcome: Closing Elastance
Description: In cmH20/mm2 - the ability of the anal canal to close after a period of stretch
Time Frame: at specific time point of measurement up to 1 hour
Measure: Mean (Standard Deviation); unit: cmH20/mm2
Arm/Group | Intra-rectal Intussusception (Oxford Groups 1 &2) | Intra-anal Intussusception (Oxford Grades 3 & 4) | Overt Rectal Prolapse (Oxford Grade 5)
Number analyzed (Participants) | 7 | 17 | 7
cmH20/mm2 | 1.52 (0.63) | 1.05 (0.46) | 0.85 (0.41)

5. Secondary Outcome: Hysteresis
Description: measured as "%" - the percentage energy dissipated during opening and closing of the anal canal at rest
Time Frame: at specific time point of measurement up to 1 hour
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Intra-rectal Intussusception (Oxford Groups 1 &2) | Intra-anal Intussusception (Oxford Grades 3 & 4) | Overt Rectal Prolapse (Oxford Grade 5)
Number analyzed (Participants) | 7 | 17 | 7
percent | 37.54 (6.32) | 39.05 (7.32) | 40.57 (11.16)

6. Secondary Outcome: Squeeze Opening Pressure
Description: the pressure (cmH2O) at whihc the anal canal opens during volunatry anal contraction
Time Frame: at specific time point of measurement up to 1 hour
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Intra-rectal Intussusception (Oxford Groups 1 &2) | Intra-anal Intussusception (Oxford Grades 3 & 4) | Overt Rectal Prolapse (Oxford Grade 5)
Number analyzed (Participants) | 7 | 17 | 7
cmH2O | 81.21 (41.46) | 82.91 (43.57) | 52.51 (33.58)

7. Secondary Outcome: Squeeze Opening Elastance
Description: the resistance of the anal canal to stretch during voluntary contraction
Time Frame: at specific time point of measurement up to 1 hour
Measure: Mean (Standard Deviation); unit: cmH20/mm2
Arm/Group | Intra-rectal Intussusception (Oxford Groups 1 &2) | Intra-anal Intussusception (Oxford Grades 3 & 4) | Overt Rectal Prolapse (Oxford Grade 5)
Number analyzed (Participants) | 7 | 17 | 7
cmH20/mm2 | 1.46 (0.31) | 1.08 (0.28) | 1.29 (0.49)

ADVERSE EVENTS:
Arm/Group | Intra-rectal Intussusception (Oxford Groups 1 &2) | Intra-anal Intussusception (Oxford Grades 3 & 4) | Overt Rectal Prolapse (Oxford Garde 5)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/17 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/17 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/17 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes